CLINICAL TRIAL: NCT01002833
Title: Comparison of Three Plasmodium Falciparum Isolates in an Experimental Human Malaria Infection
Acronym: TIP1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: L.G. Visser, MD PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: TIP1
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-02

CONDITIONS: Plasmodium Falciparum; Malaria
Keywords: Plasmodium falciparum; Malaria
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PfA (Experimental): Exposure of human volunteers to bites of mosquitoes infected with the A strain of Plasmodium falciparum
  Interventions: Biological: Exposure to Plasmodium falciparum infected mosquitoes
- PfB (Experimental): Exposure of human volunteers to bites of mosquitoes infected with the B strain of Plasmodium falciparum
  Interventions: Biological: Exposure to Plasmodium falciparum infected mosquitoes
- NF54 (Active Comparator): Exposure of human volunteers to bites of mosquitoes infected with the NF54 strain of Plasmodium falciparum
  Interventions: Biological: Exposure to Plasmodium falciparum infected mosquitoes

INTERVENTIONS:
Biological: Exposure to Plasmodium falciparum infected mosquitoes — Healthy volunteers are exposed to the bites of 5 Plasmodium falciparum infected mosquitoes

SUMMARY:
Plasmodium falciparum isolates display a wide genetic diversity with possibly different properties to induce immune responses. These properties could directly influence the ability to induce protective efficacy. Since 1998 an experimental human malaria infection model at the Radboud University Nijmegen Medical Center (RUNMC) has been very successful in answering questions with regards to immunological mechanisms of human Pf infection. To date only the NF54 strain of Pf has been deployed in this Nijmegen model. However, investigation of heterologous Pf challenge is not only highly informative for our basic understanding of induction of immune responses but also provides an essential model for protective capacity testing in the clinical development of candidate malaria vaccines. Recently, the parasite culture laboratory of the RUNMC has been able to overcome technical hurdles to produce infectious mosquitoes of two genetically different isolates from different geographical regions to increase the portfolio for Phase IIa trials. These isolates, PfA and PfB will be compared with the NF54 strain for parasitic, immunological and clinical features in humans.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 35 years healthy volunteers (males or females)
* General good health based on history and clinical examination
* Negative pregnancy test
* Use of adequate contraception for females
* All volunteers have to sign the informed consent form following proper understanding of the meaning and procedures of the study
* Volunteer agrees to inform the general practitioner and agrees to sign a request for medical information concerning contra-indications for participation in the study
* Willingness to undergo a Pf sporozoite challenge
* Agreement to stay in a hotel room close to the trial center during a part of the study (Day 5 till Day T +3)
* Reachable by mobile phone during the whole study period
* Available to attend all study visits
* Agreement to refrain from blood donation to Sanquin or for other purposes, during the course of the study
* Willingness to undergo an HIV, hepatitis B and C test
* Negative urine toxicology screening test at screening visit and day before challenge
* Willingness to take a curative regimen of Malarone®

Exclusion Criteria:

* History of malaria
* Plans to travel to endemic malaria areas during the study period
* Previous participation in any malaria vaccine study and/or positive serology for Pf
* Symptoms, physical signs and laboratory values suggestive of systemic disorders, including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric and other conditions, which could interfere with the interpretation of the study results or compromise the health of the volunteers
* History of diabetes mellitus or cancer (except basal cell carcinoma of the skin)
* History of arrhythmia's or prolonged QT-interval
* Positive family history in 1st and 2nd degree relatives for cardiac disease < 50 years old
* An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system
* Body Mass Index (BMI) below 18 or above 30 kg/m2
* Any clinically significant deviation from the normal range in biochemistry or haematology blood tests or in urine analysis
* Positive HIV, HBV or HCV tests
* Participation in any other clinical study within 30 days prior to the onset of the study
* Volunteers enrolled in any other clinical study during the study period
* Pregnant or lactating women
* Volunteers unable to give written informed consent
* Volunteers unable to be closely followed for social, geographic or psychological reasons
* Previous history of drug or alcohol abuse interfering with normal social function during a period of one year prior to enrolment in the study
* A history of psychiatric disease
* Known hypersensitivity for anti-malaria drugs
* History of severe reactions or allergy to mosquito bites
* The use of chronic immunosuppressive drugs, antibiotics, or other immune modifying drugs within three months before study onset (inhaled and topical corticosteroids are allowed) and during the study period
* Contra-indications to Malarone® including treatment taken by the volunteers that interfere with Malarone®
* Any confirmed or suspected immunosuppressive or immunodeficiency condition, including asplenia
* Co-workers of the departments of Medical Microbiology or Internal Medicine of the Radboud University Nijmegen Medical Centre or Leiden University Medical Center
* A history of sickle cell, thalassaemia trait and G6PD deficiency

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
A significant difference in kinetics of parasitemia between groups A, B and C | 35 days

SECONDARY OUTCOMES:
Immunological properties of different Plasmodium falciparum isolates | 140 days
Time to thick smear positivity between groups A, B and C | 35 days
Maximum parasitemia and duration of parasitemia as measured by PCR | 35 days
Frequency of signs and symptoms between groups A, B and C | 140 days

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] Coffeng LE, Hermsen CC, Sauerwein RW, de Vlas SJ. The Power of Malaria Vaccine Trials Using Controlled Human Malaria Infection. PLoS Comput Biol. 2017 Jan 12;13(1):e1005255. doi: 10.1371/journal.pcbi.1005255. eCollection 2017 Jan. PMID 28081133
- [Derived] Teirlinck AC, Roestenberg M, van de Vegte-Bolmer M, Scholzen A, Heinrichs MJ, Siebelink-Stoter R, Graumans W, van Gemert GJ, Teelen K, Vos MW, Nganou-Makamdop K, Borrmann S, Rozier YP, Erkens MA, Luty AJ, Hermsen CC, Sim BK, van Lieshout L, Hoffman SL, Visser LG, Sauerwein RW. NF135.C10: a new Plasmodium falciparum clone for controlled human malaria infections. J Infect Dis. 2013 Feb 15;207(4):656-60. doi: 10.1093/infdis/jis725. Epub 2012 Nov 27. PMID 23186785